CLINICAL TRIAL: NCT06990737
Title: Phase 2 Pragmatic Trial Investigating Sentinel Lymph Node Biopsy (SLNB) Efficacy and Safety in Patients With Clinically Node-Negative (cN0), High-Risk Cutaneous Squamous Cell Carcinoma (cSCC) of the Head and Neck
Brief Title: Phase 2 Pragmatic Trial of Sentinel Lymph Node Biopsy (SLNB) in Patients With Clinically Node-Negative (cN0), High-Risk Cutaneous Squamous Cell Carcinoma (cSCC) of the Head and Neck
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCDCC319
Record Dates: First submitted 2025-05-16; First posted 2025-05-25 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Cutaneous Squamous Cell Carcinoma of the Head and Neck; Clinically Node-Negative (cN0); High-Risk Cutaneous Squamous Cell Carcinoma (cSCC) of the Head and Neck
MeSH Terms: interventions — Sentinel Lymph Node Biopsy; Lymph Node Excision

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Sentinel lymph node biopsy (SLNB) + Lymphadenectomy + Adjuvant Definitive Therapy (Experimental): Participants will have SLNs excised from the affected area(s) per standard of care. Surgeon preference will dictate the order of the surgery for resecting the primary tumor. This may also coincide with a lymphadenectomy if the patient has a positive SLN. Definitive systemic therapy (e.g., radiation therapy, chemoradiation therapy) will then be administered per standard of care following surgery.
  Interventions: Procedure: Sentinel lymph node biopsy (SLNB); Procedure: Lymphadenectomy; Drug: Adjuvant Definitive Therapy

INTERVENTIONS:
Procedure: Sentinel lymph node biopsy (SLNB) — Participants will have SLNs excised from the affected area(s) per standard of care
Procedure: Lymphadenectomy — Surgeon preference will dictate the order of the surgery for resecting the primary tumor. Elective neck dissection (END) will include nodal basins based on the primary site of disease, at-risk nodal basins, and any additional dissection per the surgeon's discretion. In the event of a positive SLN, the completion neck dissection (CND) should be completed.
Drug: Adjuvant Definitive Therapy — Use of chemotherapy will depend on the specific phase of treatment and high-risk features as per standard of care and NCCN Head and Neck Cancer-Clinical Practice Guidelines in Oncology

SUMMARY:
This is a phase 2 pragmatic study at a single site that evaluates the clinical benefit of SLNB in patients with high-risk cSCC and cN0. The primary goal is to evaluate the efficacy of SLNB based on the DFS rate at 2 years post-definitive therapy.

DETAILED DESCRIPTION:
This is a phase 2 pragmatic study at a single site that evaluates the clinical benefit of SLNB in patients with high-risk cSCC and cN0. Participants must be a candidate for surgical intervention with sentinel lymph node biopsy (SLNB) and potential lymphadenectomy for treatment of cSCC. Following enrollment, participants will have preoperative lymphoscintigraphy performed before planned surgery. During surgery, participants will have SLNs excised from the affected area(s) per standard of care. Surgeon preference will dictate the order of the surgery for resecting the primary tumor. The surgeon may elect to return to the operating room for re-resection of the primary tumor to achieve a negative pathological margin. This may also coincide with a lymphadenectomy if the patient has a positive SLN. Participants will be monitored for adverse events (AEs) during and following their SLNB per institutional practices; only pre-specified AEs of interest will be documented for the study. Definitive systemic therapy (e.g., radiation therapy, chemoradiation therapy) will then be administered per standard of care following surgery.

The primary aim is to evaluate the efficacy of SLNB based on the disease-free survival (DFS) rate at 2 years post-definitive therapy compared to historical control. The patients' 2-year DFS will be analyzed using the Kaplan-Meier approach, and a one-sided log-rank test will be conducted to compare the DFS based on the historical control (50%). Secondary aims include surgical and perioperative morbidity evaluations, and efficacy evaluations assessed by 2-year local/regional control rate, 2-year overall survival, and sensitivity/ specificity of for occult nodal disease.

ELIGIBILITY:
Inclusion Criteria:

1. Must have histologically and/or biochemically confirmed head and neck cSCC
2. Must have head and neck cSCC categorized as high risk:

   1. Location in the ear or the lip,
   2. Diameter greater than 2 cm,
   3. Depth greater than 4 mm,
   4. Perineural invasion,
   5. Poorly differentiated, and/or
   6. Recurrent disease
3. Lymph-node negative (cN0) status confirmed by computed tomography (CT) imaging.
4. Candidate for surgical intervention with sentinel lymph node biopsy (SLNB) and potential lymphadenectomy for treatment of cSCC.
5. Zubrod Performance Status 0-2
6. Age ≥18 years at time of consent.
7. Provision of signed and dated informed consent form.
8. Stated willingness to comply with all study procedures and availability for the duration of the study.

Exclusion Criteria:

1. Other active cancers.
2. Definitive clinical or radiologic evidence of regional (cervical) and/or distant metastatic disease.
3. Prior non-head and neck invasive malignancy (except non-melanomatous skin cancer, including effectively treated basal cell or squamous cell skin cancer, or carcinoma in situ of the breast or cervix) unless disease free for ≥ 2 years.
4. Diagnosis of head and neck mucosal SCC.
5. Prior systemic chemotherapy for head and neck mucosal SCC; note that prior chemotherapy for a different cancer is allowable.
6. Prior radiotherapy to the head and neck that would result in overlap of radiation therapy fields.
7. Patient with severe, active co-morbidity that would preclude a lymphadenectomy.
8. Pregnant or breast-feeding persons.
9. Prior surgery involving the lateral neck, including neck dissection or gross injury to the neck that would preclude surgical dissection for this trial. Prior thyroid and central neck surgery is permissible; biopsy is permitted. Prior surgery for confirmation of tumor pathology is permitted. Note: Borderline suspicious nodes that are ≥1 cm with radiographic finding suggestive of NOT malignant should be biopsied using U/S-guided fine-needle aspirate (FNA) biopsy.
10. Underlying or documented history of hematologic malignancy (e.g., chronic lymphocytic leukemia) or other active disease capable of causing lymphadenopathy (sarcoidosis or untreated mycobacterial infection).
11. Actively receiving systemic cytotoxic chemotherapy, immunosuppressive, anti-monocyte, or immunomodulatory therapy.
12. Currently participating in another investigational therapeutic trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2031-08-01 (Estimated); Study Completion 2032-08-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | Up to 2 years post definitive therapy completion
  Defined as the time from definitive therapy to local/regional relapse, distant metastasis, or death due to any cause, whichever comes first.

SECONDARY OUTCOMES:
Number of participants experiencing surgical and perioperative morbidity | Through 30 days post-sentinel lymph node biopsy
  Assessed per the Clavien-Dindo Classification (CDC) scale 1 and a list of pre-specified complications
Local/regional control | Up to 2 years post definitive therapy completion
  Defined as the time of completing definitive therapy to any evidence of disease in the primary or regional lymph nodes based on biopsy testing or imaging.
Overall survival | Up to 2 years post definitive therapy completion
Sensitivity of sentinel lymph node biopsy for occult nodal disease | Up to 14 days post-SLNB
Specificity of sentinel lymph node biopsy for occult nodal disease | Up to 14-days post-SLNB

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Birkeland, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No